CLINICAL TRIAL: NCT05514808
Title: A Theory of Planned Behavior-based Intervention to Influence Intentions and Related Determinants for Dietary Supplement Use Among Varsity Athletes at the University of Guelph
Brief Title: An Intervention to Improve Knowledge on Dietary Supplements Among Varsity Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Responsible Party: Principal Investigator, Dalia El Khoury, Associate Professor, University of Guelph
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 22-03-003
Record Dates: First submitted 2022-08-16; First posted 2022-08-24 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Knowledge, Attitudes, Practice
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrition education intervention group (Active Comparator): Each week, participants will learn about a topic related to nutrition, health and values-based ethics of clean sport. The intervention group will also receive information on dietary supplements, their benefits and their risks. Doping and body appreciation and their links to the use of dietary supplements will also be covered in this group. The duration of the intervention is 4 weeks; 1 module to be released every week.
  Interventions: Other: Nutrition education modules
- Control group (No Intervention): No intervention to be received during the 4-week period.

INTERVENTIONS:
Other: Nutrition education modules — Nutrition education modules on sports nutrition and dietary supplements over a period of 4 weeks (1 module/week)
  Arms: Nutrition education intervention group

SUMMARY:
The aim of this project is to increase knowledge on and influence intention (and related determinants) toward the use of dietary supplements in populations at risk for doping such as university student athletes. Our objectives are to increase athletes' knowledge on dietary supplements, change their attitude, subjective norms and perceived behavioural control toward the use of these supplements, increase their body appreciation and thus increase their intention to take nutrients from diet first before considering dietary supplements. We are proposing the conceptualization, implementation, and evaluation of a nutrition education program on dietary supplements targeting varsity athletes at universities across Ontario.

Participants will be recruited from varsity teams at the University of Guelph. The intervention will be tested for validity and reliability and implemented online through Courselink modules over 4 weeks. Participants will be randomly assigned to a control or intervention group, using a randomized control trial approach. Each week, participants will learn about a topic related to nutrition, health and values-based ethics of clean sport. The intervention group will receive additional information on dietary supplements, their benefits and their risks. Doping and body appreciation and their links to the use of dietary supplements will also be covered in this group. A questionnaire assessing outcome objectives will be administered before and at the end of the intervention as well as 3 months post-intervention. Among the different components covered in the questionnaire, one section will assess knowledge on health, sports nutrition, and dietary supplements; and another will gather responses to statements reflecting the different theory of planned behaviour (TPB) cognitive constructs.

DETAILED DESCRIPTION:
High prevalence rates of dietary supplement use are consistently reported across sports disciplines in the athletic population, and this behaviour can be problematic. The use of non-prohibited dietary supplements and of doping substances are interrelated: 1) some dietary supplements are ''contaminated'' with substances prohibited by the World Anti-Doping Agency, leading to cases of inadvertent doping; and 2) supplement users are more favourable toward and more likely to engage in doping use. Many athletes derive their supplement-related information from less reliable sources as shown in a pilot study conducted by our research team on supplementation practices of varsity athletes at the University of Guelph. Also, 58.6% of those athletes mentioned wanting to become more knowledgeable about supplements. Given the findings from our pilot study, the association between dietary supplement use and risk for doping and the frequent reporting of doping rule violation among competing athletes across all types of sports in Canada, it is imperative to educate athletes about the appropriate use of dietary supplements.

The aim of this project is to increase knowledge on and influence intention (and related determinants) toward the use of dietary supplements in populations at risk for doping such as university student athletes. Our objectives are to increase athletes' knowledge on dietary supplements, change their attitude, subjective norms and perceived behavioural control toward the use of these supplements, increase their body appreciation and thus increase their intention to take nutrients from diet first before considering dietary supplements. We are proposing the conceptualization, implementation, and evaluation of a nutrition education program on dietary supplements targeting varsity athletes at universities across Ontario.

Participants will be recruited from varsity teams at the University of Guelph. The intervention will be tested for validity and reliability and implemented online through Courselink modules over 4 weeks. Participants will be randomly assigned to a control or intervention group, using a randomized control trial approach. Each week, participants will learn about a topic related to nutrition, health and values-based ethics of clean sport. The intervention group will receive additional information on dietary supplements, their benefits and their risks. Doping and body appreciation and their links to the use of dietary supplements will also be covered in this group. A questionnaire assessing outcome objectives will be administered before and at the end of the intervention as well as 3 months post-intervention. Among the different components covered in the questionnaire, one section will assess knowledge on health, sports nutrition, and dietary supplements; and another will gather responses to statements reflecting the different theory of planned behaviour (TPB) cognitive constructs.

This study will advance knowledge on dietary supplements and will support the integration of reliable educational materials on supplements into the training schedules of varsity athletes at the University of Guelph. Findings from this project will also guide the development of dietary supplement-focused educational programs at national and international levels to advance the fight against doping in sports.

ELIGIBILITY:
Inclusion Criteria:

* current University of Guelph-registered part-time or full-time student
* fluent in English
* varsity athlete

Exclusion Criteria:

* not a University of Guelph-registered student
* not fluent in English
* not a varsity athlete

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Percent of participants with correct answers to questions in the questionnaire assessing their knowledge on dietary supplements, their benefits and their risks | 4 weeks
  knowledge on dietary supplements

SECONDARY OUTCOMES:
Change in participants' theory of planned behaviour cognitive constructs with respect to the use of dietary supplements, as assessed in the questionnaire | 4 weeks
  Theory of planned behaviour cognitive constructs: intention, attitude, subjective norms, and perceived behavioural control with respect to dietary supplement use (Likert scale 1 (strongly disagree) to 5 (strongly agree))
Percent of participants with improved body image and body appreciation, as assessed in the questionnaire, in relation to the use of dietary supplements | 4 weeks
  The interaction between dietary supplement use, body image and body appreciation

CONTACTS AND LOCATIONS:
Overall Officials: Dalia El Khoury, PhD RD, Principal Investigator — University of Guelph
Locations (1):
- University of Guelph, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No